CLINICAL TRIAL: NCT03907631
Title: Elevate ASUC - Evaluating Clinical and Endoscopic Variables in Assessment, Treatment and Outcome Endpoints in Acute Severe Ulcerative Colitis
Brief Title: Multi-centre Acute Severe Ulcerative Colitis Prospective Cohort Study (Elevate ASUC)
Acronym: ELEVATE-ASUC
Status: Active, not recruiting | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 259837
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-10

CONDITIONS: Severe Ulcerative Colitis
Keywords: Rescue; Infliximab; Outcomes; Risk Stratification
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool and colonic biopsies will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Severe Ulcerative Colitis: Patients hospitalised for acute severe ulcerative colitis will be invited to participate. Participants will be treated at the discretion of their treating physicians as per standard of care. We expect some participants will undergo an endoscopic assessment, some participants will be treated with standard versus accelerated infliximab dosing, permitting comparisons, in addition to other treatment strategies.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — care decisions driven by local physicians; this is an observational cohort

SUMMARY:
Up to one third of patients with Ulcerative Colitis (UC) will require hospitalisation for severe disease (ASUC - Acute Severe Ulcerative Colitis), often within the first 12 months of diagnosis. 30-40% of people admitted to hospital with ASUC will require colectomy during the emergency admission. Investigators will develop a multi-centre prospective inception cohort of patients with ASUC with homogeneously collected detailed longitudinal clinical, endoscopic and laboratory data.

DETAILED DESCRIPTION:
ASUC can be a life threatening condition for which optimal management strategies within the acute setting are required. Such strategies remain largely ill-defined with approximately 30 - 40% of ASUC inpatient admissions requiring emergency colectomy.

Intravenous corticosteroids have been the mainstay of management during the inpatient admission but approximately 40% of this patient group will be steroid resistant. Although mortality following emergency colectomy has indeed fallen over time, it still remains as high as 10% at the 12 week marker. Patients with steroid refractory disease salvage therapy with infliximab can be considered to avoid colectomy.

Currently there are no predictive indices to identify patients needing rescue therapy. Hence health care professionals have no tools to 'personalise' care for ASUC by predicting up front which patients fail initial medical therapy and thus predict those who may benefit from rescue therapy or early surgery.

Traditionally the Truelove and Witts severity Index is used to define the clinical severity of disease on admission, but this long-standing index has yet to be validated as a predictor for the need for colectomy during the acute hospitalised phase. Similarly, endoscopic indices, including the only validated endoscopic severity score in UC (UCEIS - Ulcerative Colitis Endoscopic Index of Severity) have not been prospectively evaluated in the setting of ASUC.

Approximately 30% of ASUC patients treated with rescue anti TNF will fail to respond and require urgent colectomy. The optimal dosing regimes for rescue therapy with infliximab remains uncertain.Recently, there have been reports of increasing use of accelerated induction anti - TNF regimes in patients with ASUC (10mg/kg or shorter intervals) despite lack of clear evidence to support this practice. Randomised trial evidence for selecting patients suitable for accelerated induction regimes is not yet currently available and will require large sample size to elucidate clearly the variables that predict the need for individual dosing strategies.

Another consideration in the management of ASUC patients is the wide variability in practices among institutions and clinicians; this may potentially affect quality of care and outcomes within this cohort.

Investigators will develop a multi-centre prospective inception cohort of patients with ASUC with homogeneously collected detailed longitudinal clinical, endoscopic, laboratory and pharmacological data. This will facilitate development of risk prediction models in ASUC helping early risk stratification and supporting optimized medical and surgical algorithms in ASUC. The study will also facilitate development of a learning network in participating centres to improve quality of care.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 80 years.
* Confirmed acute severe ulcerative colitis based on modified Truelove and Witts criteria requiring hospital admission.
* Need for at least 2 days of intravenous steroids
* Able to sign consent

Exclusion Criteria:

* Crohn's disease
* Admission for elective colectomy
* Infective colitis confirmed on stool culture, assays for C. difficile or cytomegalovirus
* Pregnancy
* Inability to sign consent
* Prior colitis related surgery - pouch, stoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalised patients with Acute severe ulcerative colitis
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
In Hospital Outcomes | 30 days
  Response assessed by the following clinical care decisions based on binary outcomes: need for rescue therapy (yes = 1 or no =), need for accelerated induction (yes = 1 or no = 0), need for surgery during index admission (yes = 1 or no = 0)
Colectomy rates | 30 days
  Proportion of patients needing colectomy

SECONDARY OUTCOMES:
Long-term response to medical management | day 90 and 12 month time points
  Response assessed by the following clinical care decisions based on binary outcomes: Colectomy free survival at strategic time points (yes = 1 or no = 0)
Risk factors for need for rescue | 30
  Analysis of risk factors predicting need for rescue

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology, Hull Royal Infirmary, Hull University Teaaching Hospitals NHS Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided